CLINICAL TRIAL: NCT00060502
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo Controlled Study Evaluating the Efficacy and Safety of Anti-TNF a Monoclonal Antibody (Infliximab) to Treat Cancer-Related Cachexia in Subjects With Pancreatic Cancer.
Brief Title: A Study of the Safety and Effectiveness of Infliximab (Remicade) in Patients With Pancreatic Cancer Related Cachexia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004798
Record Dates: First submitted 2003-05-07; First posted 2003-05-08 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-04

CONDITIONS: Cachexia; Pancreatic Neoplasms
Keywords: cachexia; pancreatic cancer; infliximab; anorexia; anemia; Remicade.
MeSH Terms: conditions — Cachexia; Pancreatic Neoplasms; Anorexia; Anemia | interventions — Infliximab; Gemcitabine

INTERVENTIONS:
Drug: Infliximab; Gemcitabine

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of infliximab, the active ingredient in Remicade, for the treatment of cachexia in pancreatic cancer patients who are receiving chemotherapy with gemcitabine.

DETAILED DESCRIPTION:
Cachexia is a condition that occurs in cancer patients and other chronically ill patients and is characterized by rapid loss of fatty tissue and skeletal muscle. The key feature of this condition is weight loss, but other symptoms, such as anorexia (loss of appetite), fatigue, vomiting and anemia (low numbers of red blood cells) may also occur.The purpose of this study is to evaluate the effectiveness and safety of infliximab, the active ingredient in Remicade, for the treatment of cachexia in pancreatic cancer patients who are receiving chemotherapy with gemcitabine. In cycle 1 (8wks), patients will receive weekly infusions of gemcitabine from wk 0 to 6 and infusions of infliximab or placebo at wks 0, 2, and 4. For additional cycles, patients will receive an infusion of gemcitabine for the first 3wks and infliximab or placebo at wk 0 of each 4 wk cycle for a maximum of 5 cycles. Patients with stable disease may receive extended dosing if qualified.Safety evaluations will be performed at specified intervals throughout the study and will consist of laboratory tests, vital signs (such as blood pressure), physical examinations and the occurrence and severity of adverse events as well as other study specific procedures. In cycle 1 (8wks), patients will receive weekly infusions of gemcitabine from wk 0 to 6 and infusions of infliximab or placebo at wks 0, 2, and 4. For additional cycles, patients will receive an infusion of gemcitabine for the first 3wks and infliximab or placebo at wk 0 of each 4 wk cycle for a maximum of 5 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have documented diagnosis of pancreatic cancer that is newly diagnosed
* Patients must have documented loss of >=10% body weight compared to weight prior to diagnosis, or >=5% weight loss within 90 days prior to randomization
* Patients must have Karnofsky performance status of 70 to 100
* eligible according to country specific tuberculosis (TB) screening rules.

Exclusion Criteria:

* Patients must not have received any previous chemotherapy, biologic therapy or radiation therapy for pancreatic cancer
* Patients must not have a history or current evidence of active TB, skin test or screening evidence of latent TB, or history of treated TB, active or latent
* Patients must not have evidence or history of congestive heart failure
* Patients must not have any opportunistic infection within 6 months prior to screening
* Patients must not be pregnant, nursing or planning pregnancy
* Patients must not have ongoing use of tube feedings or TPN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2003-04; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Change in Lean Body Mass (LBM) from baseline to the end of first cycle, as measured by bioelectrical impedance analysis (BIA).

SECONDARY OUTCOMES:
Change in 6-minute walk test distance from baseline to the end of the first cycle; Safety, Karnofsky performance status; Survival.

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Result] Wiedenmann B, Malfertheiner P, Friess H, Ritch P, Arseneau J, Mantovani G, Caprioni F, Van Cutsem E, Richel D, DeWitte M, Qi M, Robinson D Jr, Zhong B, De Boer C, Lu JD, Prabhakar U, Corringham R, Von Hoff D. A multicenter, phase II study of infliximab plus gemcitabine in pancreatic cancer cachexia. J Support Oncol. 2008 Jan;6(1):18-25. PMID 18257397
- See also: A Phase II, Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of Anti-TNFa Monoclonal Antibody (Infliximab) to Treat Cancer-related Cachexia in Subjects with Pancreatic Cancer — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=156&filename=CR004798_CSR.pdf